CLINICAL TRIAL: NCT02828475
Title: Pilot Study for a Clinical Analytical Platform for Surgical Outcomes
Brief Title: CALYPSO Pilot Study: Machine Learning Based Predictions of Surgical Complications
Acronym: CALYPSO
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00072563
Record Dates: First submitted 2016-07-07; First posted 2016-07-11 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-01

CONDITIONS: Complication of Surgical Procedure; Postoperative Infection
MeSH Terms: interventions — thiacloprid; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CALYPSO-augmented: Patients' postoperative care will be augmented with the CALYPSO platform.
  Interventions: Other: CALYPSO; Behavioral: Standard Care
- Historical Control: Patients' postoperative care was performed using standard practice, before adopting the CALYPSO platform
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Other: CALYPSO — Software platform of machine-learning based predictive models of surgical complication.
  Groups: CALYPSO-augmented
Behavioral: Standard Care — Previous standard of care based on surgeon judgement alone.

SUMMARY:
This is a pilot study of surgical patients whose postoperative care will be augmented with a personalized risk prediction platform (CALYPSO app).

DETAILED DESCRIPTION:
CALYPSO is a software platform that uses machine learning techniques to create personalized risk predictions for postoperative complications. Individual risk factors are then linked to best-practice interventions tailored to the individual patient. The investigator aims to test the hypothesis that using CALYPSO-augmented postoperative care will reduce complication rates in patients undergoing elective general surgery. Subjects undergoing surgery will be assigned to the CALYPSO intervention in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Undergoing elective surgery
* Undergoing high risk colon, rectal, pancreas, gastric surgery with predicted length of stay greater or equal to 3 days

Exclusion Criteria:

* Surgeries with less than 3 days of anticipated length of stay (e.g. stoma takedown)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing high risk general and oncologic abdominal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Thirty Day Overall Complications | 30 days after surgery

SECONDARY OUTCOMES:
Thirty Day Mortality | 30 days after surgery
Wound Complications | 30 days after surgery
  Includes superficial, deep, organ space infections, and wound dehiscence
Cardiac Complications | 30 days after surgery
  includes myocardial infarction, cardiac arrest
Respiratory Complications | 30 days after surgery
  includes unplanned reintubation, pneumonia, failure to wean from ventilator >48 hours after surgery
Thrombotic complications | 30 days after surgery
  includes deep vein thrombosis, pulmonary emobolism
Renal Complications | 30 days after surgery
  includes acute renal failure, renal failure requiring dialysis
urinary tract infections | 30 days after surgery
Neurologic complications | 30 days after surgery
  includes stroke, peripheral nerve injury, coma
Septic complications | 30 days after surgery
  includes sepsis and septic shock
Unplanned reoperation | 30 days after surgery
unplanned readmission | 30 days after surgery
bleeding complications | up to 72 hours after surgery
  needing at least 1 unit of pRBC

CONTACTS AND LOCATIONS:
Overall Officials: Zhifei Sun, MD, Study Director — Duke University Department of Surgery
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No